CLINICAL TRIAL: NCT06057363
Title: Volumetric and Clinical Evaluation of Peri-implant Soft Tissue Augmentation in Different Sites After Laser-aided Pouch Roll Technique: a Prospective Study
Brief Title: Volumetric Evaluation of Gingival Augmentation Around Dental Implants
Status: Completed | Type: Observational
Sponsor: Odontostomatologic Laser Therapy Center, Florence, Italy (Other)
Collaborators: University of Florence (Other)
Responsible Party: Sponsor
Other Study IDs: 20546-oss
Record Dates: First submitted 2023-09-13; First posted 2023-09-28 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Atrophy of Gingiva
Keywords: dental implants; roll flap; gingival augmentation; volume changes; linear dimensional changes; clinical periodontal parameters; patient-reported outcomes
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients requiring vestibular soft tissue augmentation at implant sites: The present study was planned as prospective analysis with 12-month follow-up. It enrolled 12 partially edentulous patients (mean age 62; range 42-86) requiring vestibular soft tissue augmentation at implant sites in second-stage surgery because of mild horizontal ridge deficiency. As a whole, 16 implants were placed (8 single, 4 dual).
  Interventions: Other: volumetric evaluation of gingival augmentation around dental implants

INTERVENTIONS:
Other: volumetric evaluation of gingival augmentation around dental implants — objective volumetric and clinical assesment of vestibular gingival soft tissues changes upon treatment with laser-aided pouch roll augmentation technique and implant placement over a 12-month follow-up

SUMMARY:
The goal of this observational prospective study is to objectively assess the dimensional (volume & linear variance) and clinical changes of vestibular gingival soft tissues upon treatment with laser-aided pouch roll augmentation technique and implant placement over a 12-month follow-up. Twelve patients with 16 mild horizontal ridge deficiencies in different edentulous sites scheduled for implant placement were enrolled. Digital impressions were taken with an intra-oral laser scanner and software and analyzed before (day 0) and 12 months after laser-aided pouch roll augmentation surgery. The digital files were converted to STL format and superimposed to assess peri-implant volumetric and linear dimensional variations in selected regions of interest (ROI) by a 3D analysis software. Operator-assessed clinical periodontal parameters (probing depth PD, bleeding on probing BoP, plaque index PI) were recorded. Patient-reported outcome (pain, discomfort, treatment liking) and aesthetic result were evaluated by administration of appropriate questionnaires.

DETAILED DESCRIPTION:
Introduction Adequate soft tissue thickness at the vestibular aspect of dental implants are crucial for satisfactory implant engraftment and aesthetic outcome. To pursue this objective, numerous surgical procedures have been adopted to augment the peri-implant gingiva, including autologous soft tissue grafting, xenogeneic collagen matrix, acellular dermal matrix, and roll/pedicle flap techniques: however, the available data do not suffice to clearly indicate which technique yields the best results.

The pouch roll techniques, originally proposed by Abrams in 1980 and subsequently improved, are particularly effective because they maintain vascularity of the grafted flap, which greatly facilitates its survival. Most of these procedures use a scalpel to shape the flap and remove the keratinized epithelial layer, but this conventional pouch roll technique is hampered by the fact that flap thickness must be no less than 3 mm and it is very difficult to perform hand scalpel gingival de-epithelization of the without damaging the underlying connective tissue, thereby causing bleeding and predisposing to scarring in the long term. More recently, laser-aided epithelial photoablation has been proposed as a possible solution to these issues. In fact, diode laser operating at 810 nm wavelength (λ) has been successfully used for selective de-epithelialization for several periodontal therapy purposes, e.g. palatal grafts for gingival recession defects, gingival hyperpigmentation, intra/extra pocket decontamination in chronic periodontitis and placement to second-stage surgery for buried implant exposure. Laser photoablation offers several advantages, namely excellent hemostasis that results in a dry surgical field and better view of the operative field, tissue surface sterilization and shallow penetration limited to the gingival epithelium with minimal injury and inflammation of the underlying lamina propria. On this ground, the investigators successfully combined diode laser photoablation (λ 810 nm) to conventional roll flap technique for mild vestibular ridge deficiencies: in a preliminary, limited series of patients (n=3) this improved method resulted in fast healing, satisfactory clinical and aesthetic results, rapid prosthetic restoration and no need for local or systemic analgesics. The present study aims on one hand at expanding the case series to consolidate the preliminary findings, on the other hand at evaluating another key clinical outcome parameter of this laser-aided roll flap procedure, namely the actual, objective gingival soft tissue augmentation over time. To this purpose, the volume of the treated regions, acquired by a digital intra-oral scanning, was measured and analyzed by appropriate 3D software and compared before roll flap surgery and implant placement and upon 12-month follow-up. Post-operative discomfort and aesthetic satisfaction of the patients were also assessed.

Material and methods

Volumetric measurements and analysis - Volume changes of the vestibular gingiva before and after the laser-aided roll-flap augmentation were evaluated and compared on digital intra-oral scanning impressions taken with an intra-oral scanner (Dentsply Syrona, Rome, Italy) and 3D reconstruction software (Exocad, Darmstadt, Germany). To reduce possible deviations and ensure higher accuracy of 3D analysis, quadrant instead of full-arch scans were recorded. These were converted to standard tessellation language (STL) format. Pre and post-operative STL files were collected, aligned and superimposed by selecting 10 reproducible anatomical points as landmarks prior to be analyzed with an appropriate software (Rhyno3D, Washington DC, USA). This software allowed: i) to demarcate an exact 3D region of interest (ROI), ii) to superimpose the same ROI taken at 2 time points, i.e. before surgery (day 0) and at 12-month follow-up, while to measure the volume of the 2 corresponding ROI and to objectively assess their differences at the different time points. Each selected ROI corresponded to a single or multiple implant site. According to previous studies, ROI in the single implant sites was demarcated on the vestibular gingival aspect using the following criteria:

1. gingiva-to-implant margin (or coronal gingival ridge, if before implant placement) as horizontal coronal border;
2. muco-gingival junction as horizontal apical border;
3. two vertical lines, 2 mm aside the surgical flap incision and corresponding to the mid-point of the interdental papillas, as mesial and distal borders.

Due to individual variations in oral anatomy, ROI were obviously different among the patients, but substantially identical in the same patient at successive time points. The software was set to a spatial resolution of ±50 nm between the STL files: in this way, negligible or no variations <50 nm in the merged STL file appeared green in a visual pseudo-color range. To assess reproducibility of the method, a trained blinded examiner (M.P.), performed 2 measurements at 1-week interval: intra-class correlation coefficient was 0.87 (95% CI 0.82-0.91).

In each patient, the 2 ROI volumes (cubic mm) measured at day 0 and 12 months were compared to evaluate the changes of the vestibular gingival soft tissue over time. Exocad software also allowed to determine the linear dimensional changes (LD), i.e. the linear distance (mm) between the 2 ROI surfaces measured at 1, 3 and 5 mm along a vertical midline traced between the gingival free margin and the muco-gingival junction, as previously reported.

Clinical peri-implant parameters and calibration - At 12 months, a trained and blinded examiner (L.L.) evaluated PD and BoP (within 30 s after probing) at 6 sites per implant (3 buccal, 3 palatal) and PI (yes/no, 4 sites per implant), using a conventional manual periodontal probe (PCP15, Hu-Friedy, Milan, Italy) with about a 0.3 N force. Operator calibration was considered satisfactory when the percent fitting between the first and second measurements taken at a 24-h gap was ≥ 90%.

Primary outcome variables

1. Objectively measurable volumetric changes (cubic mm) of the ROI regions between day 0 and 12 months.
2. Objectively measurable linear dimensional changes (LD, mm) of the ROI regions between day 0 and 12 months;

Secondary outcome variables

1. Changes in periodontal probing depth PD (mm)
2. Changes in periodontal bleeding on probing BoP (yes/no),
3. Changes in plaque index PI (yes/no)
4. Subjective perception of discomfort and pain during surgery and the post-operative period, semi-quantitatively assessed by Visual Analogue Scale (VAS) questionnaires administered 5 h after surgery and each morning for the next 7 days (score: 0,no pain to 10,extremely painful);
5. analgesics taken (number);
6. willingness to undergo the same treatment again (yes/no).
7. Color and texture differences between peri-implant and natural gingiva at 12 months, subjectively evaluated by the patients at a mirror from speaking distance (visible/not visible).

Operators - Laser-aided roll-flap technique was performed by a dental practitioner (M.G) with long-lasting expertise in periodontal surgery, implant dentistry and use of dental laser technology.

Surgical treatments - The delivered laser-aided roll flap technique was performed as previously described. It consisted in the following steps:

1. De-epithelialization of a vestibular gingival area, 2 mm larger than the cover screw diameter, using a λ 810-nm diode GaAlAs laser (4x4 Dental Laser System, General Project Ltd., Montespertoli, Florence, Italy) equipped with a ∅ 600-μm optical fiber and set as follows: pulse mode, frequency 8,000 Hz, pulse energy 69 μJ, pulse duration 18 μs, corresponding to 0.6 W
2. mean power (peak 3.8 W) and 40 J/square cm irradiation energy. Photoablation was performed in fiber tip contact mode at a constant speed of about 2.5 mm/s under airflow cooling and thermographic feedback to prevent tissue over-heating and damage. The procedure was made under a high-resolution stereomicroscope (Extaro 300, Zeiss, Milan, Italy).
3. Full-thickness U-shaped incision of the photoablated mucosa was made with the same λ 810-nm diode laser set at pulse energy 22 μJ, peak power 3.14 W, frequency 20 kHz, pulse width 7 μs, in contact mode and equipped with a ∅ 300-μm optical fiber. The incision margins were extended to the vestibular gingiva for 2 to 3 mm to facilitate flap displacement.
4. Elevation and rolling of the full-thickness flap into a vestibular pouch, no surgical sutures.
5. Relieve or remove any soft tissue or bone interferences by adjusting the abutment or the tissues.
6. Connection of titanium abutments or healing abutment to the implants. Overall time of the surgical procedure was measured, starting from the end of local anesthesia to connection of titanium abutment.

Post-surgical instructions and prosthetic treatments - No local or systemic antibiotics, mouthwashes or toothpastes containing triclosan, chlorhexidine, or other disinfectants were prescribed. The patients were instructed to avoid brushing of the treated zone for about 6 hours from surgery and then to perform normal oral hygiene.

Prosthetic treatment including the application of a temporary crown and the final rehabilitation was performed according to a standard treatment plan.

Statistical analysis - This was performed with Prism5 software (GraphPad, Boston, MA, USA). The ROI of each treated implant/tooth site was taken as unit of analysis. Differences in ROI volumes (mean ±SEM) measured before the treatment (day 0) and at 12-month follow-up were analysed statistically by Student's t test for paired values. A p value ≤0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Self-reported smoking habits >10 cigarettes/day.
3. Full-mouth plaque score and full-mouth bleeding score ≤15%, measured at four sites per tooth.
4. Need for aesthetic and/or functional soft tissue augmentation in single or multiple implant sites at the upper and/or lower quadrants.

Exclusion Criteria:

1. Diseases affecting connective tissue metabolism.
2. Uncontrolled diabetes (glycated hemoglobin HbA1c >7).
3. Pregnant or lactating women.
4. Untreated periodontal disease.
5. Heavy gingival pigmentation (grade 3 Dummet Oral Pigmentation Index) requiring substantially different photoablative laser settings

Ages: 42 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 12 partially edentulous patients (mean age 62; range 42-86; 9 males/5 females) requiring vestibular soft tissue augmentation at implant sites in second-stage surgery because of mild horizontal ridge deficiency were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Objectively measurable volume changes of the vestibular gingiva | 12 months
  Assessment of peri-implant volumetric variations (cubic mm) in selected regions of interest (ROI) of the vestibular gingiva by a 3D analysis software
Objectively measurable linear dimensional (LD) changes of the vestibular gingiva | 12 months
  Assessment of peri-implant linear dimensional variations (mm) at 3 vertical points (1,3,5 mm form the free margin) in selected regions of interest (ROI) of the vestibular gingiva by a 3D analysis software

SECONDARY OUTCOMES:
Changes in periodontal probing depth PD (mm) | 12 months
  Operator-assessed periodontal probing depth (PD), in mm
Changes in periodontal bleeding on probing BoP | 12 months
  Operator-assessed periodontal bleeding on probing (BoP) within 30 s, 6 sites per implant (yes/no)
Changes in periodontal plaque index PI | 12 months
  Operator-assessed periodontal plaque index, 4 sites per implant (yes/no)
Subjective perception of discomfort and pain during surgery and the post-operative period | 7 days
  Patient-reported perception of discomfort and pain during surgery and the post-operative period, semi-quantitatively assessed by Visual Analogue Scale (VAS) questionnaires administered 5 h after surgery and each morning for the next 7 days (score: 0,no pain to 10,extremely painful)
Analgesics taken | 7 days
  Patient-reported No. of pills of analgesics taken after surgery and in the next days
Treatment liking | 7 days
  Patient-reported willingness to undergo the same treatment again (yes/no)
Gingival color and texture appearance | 12 months
  Patient-reported color and texture differences between peri-implant and natural gingiva, subjectively evaluated at a mirror from speaking distance (visible/not visible).

CONTACTS AND LOCATIONS:
Overall Officials: Marco Giannelli, MD, Principal Investigator — Odontostomatologic Laser Therapy Center
Locations (1):
- Odontostomatologic Laser Therapy Center, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams L. Augmentation of the deformed residual edentulous ridge for fixed prosthesis. Compend Contin Educ Gen Dent. 1980 May-Jun;1(3):205-13. No abstract available. PMID 6950834
- [Background] Bassetti RG, Stahli A, Bassetti MA, Sculean A. Soft tissue augmentation around osseointegrated and uncovered dental implants: a systematic review. Clin Oral Investig. 2017 Jan;21(1):53-70. doi: 10.1007/s00784-016-2007-9. Epub 2016 Nov 21. PMID 27873018
- [Background] El-Kholey KE. Efficacy and safety of a diode laser in second-stage implant surgery: a comparative study. Int J Oral Maxillofac Surg. 2014 May;43(5):633-8. doi: 10.1016/j.ijom.2013.10.003. Epub 2013 Nov 7. PMID 24210453
- [Background] Fons-Badal C, Alonso Perez-Barquero J, Martinez-Martinez N, Faus-Lopez J, Fons-Font A, Agustin-Panadero R. A novel, fully digital approach to quantifying volume gain after soft tissue graft surgery. A pilot study. J Clin Periodontol. 2020 May;47(5):614-620. doi: 10.1111/jcpe.13235. Epub 2020 Mar 12. PMID 31860133
- [Background] Fornaini C, Merigo E, Vescovi P, Bonanini M, Antonietti W, Leoci L, Lagori G, Meleti M. Different laser wavelengths comparison in the second-stage implant surgery: an ex vivo study. Lasers Med Sci. 2015 Aug;30(6):1631-9. doi: 10.1007/s10103-014-1623-3. Epub 2014 Jul 3. PMID 24989333
- [Background] Giannelli M, Formigli L, Bani D. Comparative evaluation of photoablative efficacy of erbium: yttrium-aluminium-garnet and diode laser for the treatment of gingival hyperpigmentation. A randomized split-mouth clinical trial. J Periodontol. 2014 Apr;85(4):554-61. doi: 10.1902/jop.2013.130219. Epub 2013 Jul 4. PMID 23826649
- [Background] Giannelli M, Formigli L, Lorenzini L, Bani D. Combined photoablative and photodynamic diode laser therapy as an adjunct to non-surgical periodontal treatment: a randomized split-mouth clinical trial. J Clin Periodontol. 2012 Oct;39(10):962-70. doi: 10.1111/j.1600-051X.2012.01925.x. Epub 2012 Jul 27. PMID 22834932
- [Background] Gonzalez-Martin O, Veltri M, Moraguez O, Belser UC. Quantitative three-dimensional methodology to assess volumetric and profilometric outcome of subepithelial connective tissue grafting at pontic sites: a prospective pilot study. Int J Periodontics Restorative Dent. 2014 Sep-Oct;34(5):673-9. doi: 10.11607/prd.1808. PMID 25171038
- [Background] Ozcelik O, Seydaoglu G, Haytac CM. Diode laser for harvesting de-epithelialized palatal graft in the treatment of gingival recession defects: a randomized clinical trial. J Clin Periodontol. 2016 Jan;43(1):63-71. doi: 10.1111/jcpe.12487. Epub 2016 Jan 21. PMID 26660000
- [Background] Park SH, Wang HL. Pouch roll technique for implant soft tissue augmentation: a variation of the modified roll technique. Int J Periodontics Restorative Dent. 2012 Jun;32(3):e116-21. PMID 22408781
- [Background] Parvini P, Galarraga-Vinueza ME, Obreja K, Magini RS, Sader R, Schwarz F. Prospective study assessing three-dimensional changes of mucosal healing following soft tissue augmentation using free gingival grafts. J Periodontol. 2021 Mar;92(3):400-408. doi: 10.1002/JPER.19-0640. Epub 2020 Aug 21. PMID 33448379
- [Background] Schmidt A, Klussmann L, Wostmann B, Schlenz MA. Accuracy of Digital and Conventional Full-Arch Impressions in Patients: An Update. J Clin Med. 2020 Mar 4;9(3):688. doi: 10.3390/jcm9030688. PMID 32143433
- [Background] Tavelli L, Barootchi S, Majzoub J, Siqueira R, Mendonca G, Wang HL. Volumetric changes at implant sites: A systematic appraisal of traditional methods and optical scanning-based digital technologies. J Clin Periodontol. 2021 Feb;48(2):315-334. doi: 10.1111/jcpe.13401. Epub 2020 Nov 18. PMID 33151586
- [Background] Thoma DS, Naenni N, Figuero E, Hammerle CHF, Schwarz F, Jung RE, Sanz-Sanchez I. Effects of soft tissue augmentation procedures on peri-implant health or disease: A systematic review and meta-analysis. Clin Oral Implants Res. 2018 Mar;29 Suppl 15:32-49. doi: 10.1111/clr.13114. PMID 29498129
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014 Dec;12(12):1495-9. doi: 10.1016/j.ijsu.2014.07.013. Epub 2014 Jul 18. PMID 25046131